CLINICAL TRIAL: NCT00398437
Title: Role of Gadolinium Enhanced Brain Magnetic Resonance in the Follow Up of Metastatic Breast Cancer Patients Overexpressing HER2 Neu. A Randomized Prospective Study
Brief Title: Magnetic Resonance Imaging for the Early Detection of CNS Metastases in Women With Stage IV Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: IJB-HER2-NEU-CE-1384; CDR0000516004 (Registry Identifier: PDQ (Physician Data Query)); EU-20655; EUDRACT-2006-001591
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-03

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — Trastuzumab; Drug Therapy; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Biological: trastuzumab
Drug: chemotherapy
Procedure: magnetic resonance imaging

SUMMARY:
RATIONALE: Diagnostic procedures, such as magnetic resonance imaging (MRI), may help doctors find CNS metastases and plan treatment.

PURPOSE: This randomized clinical trial is studying how well MRI finds CNS metastases in women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine survival (without neurological symptoms due to CNS metastases) in women with HER2/neu-overexpressing stage IV breast cancer who undergo gadolinium-enhanced magnetic resonance imaging (MRI) of the brain once every 4 months vs once every 12 months for early detection of CNS metastases.

Secondary

* Determine the total number of therapeutic procedures (i.e., gamma-knife, radiotherapy, or surgery) required for the treatment of brain metastases in these women.
* Determine the total number of hospitalization days required in these women.
* Determine the overall survival of these women.
* Evaluate a cross-platform, manufacturer-independent MRI technique for diagnosis of brain metastases that could be used in future studies in the IRIS and ULB-Canceropôle networks.
* Compare 2D-SE vs 3D-GE thin sections methods for post-contrast brain imaging in these women.

OUTLINE: This is a prospective, randomized study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients undergo gadolinium-enhanced magnetic resonance imaging (MRI) of the brain at baseline (to exclude CNS involvement) and then once every 4 months (or earlier if symptoms possibly related to CNS involvement develop) in the absence of the development of CNS metastases.
* Arm II: Patients undergo gadolinium-enhanced MRI of the brain at baseline (to exclude CNS involvement) and then once every 12 months (or earlier if symptoms possibly related to CNS involvement develop) in the absence of the development of CNS metastases.

Patients complete neurological symptoms questionnaires at baseline, every 6 weeks during study intervention, and at the completion of the study.

PROJECTED ACCRUAL: A total of 96 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage IV disease
* HER2/neu-overexpression (3+ by immunohistochemistry AND/OR gene amplification by fluorescence in situ hybridization)
* Undergoing treatment with trastuzumab (Herceptin®) (alone or together with chemotherapy) once weekly or 3 times weekly AND has achieved responding or stable disease for ≥ 12 weeks
* No CNS metastases (i.e., brain parenchymal lesions and/or leptomeningeal carcinomatosis)
* No uncontrolled metastatic disease at study entry
* Hormone receptor status

  * Not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Karnofsky performance status 70-100%
* No contraindication to MRI scan

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Survival without neurological symptoms due to brain metastasis and/or leptomeningeal involvement

SECONDARY OUTCOMES:
Total number of therapeutic procedures (i.e., gamma-knife, radiotherapy, or surgery) required for the treatment of brain metastases
Total number of hospitalization days required
Overall survival
Cross-platform, manufacturer-independent magnetic resonance imaging technique for diagnosis of brain metastases
Comparative evaluation of 2D-SE vs 3D-GE thin sections methods for post-contrast brain imaging

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Lebrun, MD, Study Chair — Jules Bordet Institute
Locations (3):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Centre Hospitalier Etterbeek Ixelles, Brussels